CLINICAL TRIAL: NCT02522351
Title: Reduction of Aspiration Through Cohesive Thin Liquids (CTL) in Patients With Mild Oropharyngeal Dysphagia Due to Ischemic/Hemorrhagic Cerebral Cause (Stroke)
Brief Title: Reduction of Aspiration Through Cohesive Thin Liquids (CTL) in Patients With Mild Oropharyngeal Dysphagia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 13.21. NRC
Record Dates: First submitted 2015-07-13; First posted 2015-08-13 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Dysphagia; Stroke
MeSH Terms: conditions — Deglutition Disorders; Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Thicken Up Clear concentration 1 (Active Comparator): Thicken Up Clear at concentration 1
  Interventions: Other: Cereal extract concentration 1; Other: Cereal extract concentration 2; Other: Cereal extract concentration 3; Other: Thicken up clear concentration 2; Other: Thicken up clear concentration 3
- Thicken Up Clear concentration 2 (Active Comparator): Thicken Up Clear at concentration 2
  Interventions: Other: Cereal extract concentration 1; Other: Cereal extract concentration 2; Other: Cereal extract concentration 3; Other: Thicken up clear concentration 1; Other: Thicken up clear concentration 3
- Thicken Up Clear concentration 3 (Active Comparator): Thicken Up Clear at concentration 3
  Interventions: Other: Cereal extract concentration 1; Other: Cereal extract concentration 2; Other: Cereal extract concentration 3; Other: Thicken up clear concentration 1; Other: Thicken up clear concentration 2
- Cereal extract concentration 1 (Experimental): Cereal extract at concentration 1
  Interventions: Other: Cereal extract concentration 2; Other: Cereal extract concentration 3; Other: Thicken up clear concentration 1; Other: Thicken up clear concentration 2; Other: Thicken up clear concentration 3
- Cereal extract concentration 2 (Experimental): Cereal extract at concentration 2
  Interventions: Other: Cereal extract concentration 1; Other: Cereal extract concentration 3; Other: Thicken up clear concentration 1; Other: Thicken up clear concentration 2; Other: Thicken up clear concentration 3
- Cereal extract concentration 3 (Experimental): Cereal extract at concentration 3
  Interventions: Other: Cereal extract concentration 1; Other: Cereal extract concentration 2; Other: Thicken up clear concentration 1; Other: Thicken up clear concentration 2; Other: Thicken up clear concentration 3

INTERVENTIONS:
Other: Cereal extract concentration 1 — Cereal extract will be given to see the effect on penetration and aspiration in patients with dysphagia problem
  Arms: Cereal extract concentration 2; Cereal extract concentration 3; Thicken Up Clear concentration 1; Thicken Up Clear concentration 2; Thicken Up Clear concentration 3
Other: Cereal extract concentration 2 — Cereal extract will be given to see the effect on penetration and aspiration in patients with dysphagia problem
  Arms: Cereal extract concentration 1; Cereal extract concentration 3; Thicken Up Clear concentration 1; Thicken Up Clear concentration 2; Thicken Up Clear concentration 3
Other: Cereal extract concentration 3 — Cereal extract will be given to see the effect on penetration and aspiration in patients with dysphagia problem
  Arms: Cereal extract concentration 1; Cereal extract concentration 2; Thicken Up Clear concentration 1; Thicken Up Clear concentration 2; Thicken Up Clear concentration 3
Other: Thicken up clear concentration 1 — Thicken up clear will be given to see the effect on penetration and aspiration in patients with dysphagia problem
  Arms: Cereal extract concentration 1; Cereal extract concentration 2; Cereal extract concentration 3; Thicken Up Clear concentration 2; Thicken Up Clear concentration 3
Other: Thicken up clear concentration 2 — Thicken up clear will be given to see the effect on penetration and aspiration in patients with dysphagia problem
  Arms: Cereal extract concentration 1; Cereal extract concentration 2; Cereal extract concentration 3; Thicken Up Clear concentration 1; Thicken Up Clear concentration 3
Other: Thicken up clear concentration 3 — Thicken up clear will be given to see the effect on penetration and aspiration in patients with dysphagia problem
  Arms: Cereal extract concentration 1; Cereal extract concentration 2; Cereal extract concentration 3; Thicken Up Clear concentration 1; Thicken Up Clear concentration 2

SUMMARY:
The aim of the trial is to identify any systematic effect of cohesiveness on the efficacy of swallowing in patients having dysphagia problems.

DETAILED DESCRIPTION:
This trial will be a double blind, randomized, crossover, controlled, and interventional trial. Each subject will test 6 study samples in a randomized order at 5 mL of volume first then at 10 mL (12 samples maximum). The trial will last a maximum of one hour (a single study visit).

The total sample size is 47 enrolled subjects, 33 subjects completed. Patients will be females and males aged between 18 and 85 years with mild proven dysphagia.

ELIGIBILITY:
Inclusion Criteria:

1. Mild dysphagia as defined by a score between 3 and 5 on the Dysphagia Outcome and Severity Scale
2. Patients aged between 18 and 85 years
3. Ischemic/hemorrhagic cerebral cause (stroke)
4. Able to understand French (oral and written)
5. Cognitive capacity enough to understand study procedures
6. Having health insurance (which in France is " social security")
7. Having signed the consent form.

Exclusion Criteria:

1. Any swallowing trouble not resulting from the current stroke
2. History of inhalation pneumopathy, i.e. any pulmonary inflammation linked to the path of a solid or liquid food in the respiratory system
3. Any physician diagnosed psychiatric illness
4. Patient with a digestive fistula
5. Any physician diagnosed food allergy
6. Any known allergy to barium or any compound of the contrast product
7. Confirmed or suspected perforated and occlusive syndrome
8. Pregnant or lactating women
9. Major respiratory disease needing oxygen (chronic respiratory insufficiency)
10. Subject who cannot be expected to comply with the study procedures, including consuming the test products.
11. Currently participating or having participated in another clinical trial during the month preceding the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Identification of any systematic effect of cohesiveness on the efficacy of swallowing in dysphagic patients according to Rosenbek's Penetration-Aspiration Score (PAS) using videofluoroscopy | During the ingestion (videofluoroscopy), maximum during one hour.
  The PAS score across each bolus (5 mL and 10 mL)

SECONDARY OUTCOMES:
Swallowing safety- prevalence of penetration | During the ingestion (videofluoroscopy), maximum during one hour.
  The prevalence of penetration in the population according to Rosenbek's PAS (score of 2-5) assessed using videofluoroscopy
Swallowing safety- prevalence of aspiration | During the ingestion (videofluoroscopy), maximum during one hour.
  The prevalence of aspiration in the population according to Rosenbek's PAS (score of 6-8) assessed using videofluoroscopy
Swallowing function- Amount/volume of oral and pharyngeal residues | During the ingestion (videofluoroscopy), maximum during one hour.
  The amount/volume of oral and pharyngeal residues assessed using videofluoroscopy
Swallowing function- Prevalence of subjects with oral and pharyngeal residues | During the ingestion (videofluoroscopy), maximum during one hour.
  The prevalence of subjects of oral and pharyngeal residues assessed using videofluoroscopy
Swallowing function- Oral transit time (OTT, time between tongue tip elevation and arrival of the bolus at the ramus of the mandible) | During the ingestion (videofluoroscopy), maximum during one hour.
  Oral transit time (OTT, time between tongue tip elevation and arrival of the bolus at the ramus of the mandible)
Swallowing function- Swallow response time (SRT, time between arrival of the bolus at the ramus of the mandible and pharyngeal phases of swallowing) | During the ingestion (videofluoroscopy), maximum during one hour.
  Swallow response time (SRT, time between arrival of the bolus at the ramus of the mandible and pharyngeal phases of swallowing)
Swallowing function- Pharyngeal transit time (PTT, time between arrival of the bolus at the ramus of the mandible and the tail of the bolus passing through the upper esophageal sphincter) | During the ingestion (videofluoroscopy), maximum during one hour.
  Pharyngeal transit time (PTT, time between arrival of the bolus at the ramus of the mandible and the tail of the bolus passing through the upper esophageal sphincter)
Swallowing function- Time to upper esophageal sphincter opening (UESO, time between tongue tip elevation and opening of the upper esophageal sphincter) | During the ingestion (videofluoroscopy), maximum during one hour.
  Time to upper esophageal sphincter opening (UESO, time between tongue tip elevation and opening of the upper esophageal sphincter)
Swallowing function-Time to laryngeal vestibule opening (LVO, time between tongue tip elevation and pharyngeal phases of swallowing) | During the ingestion (videofluoroscopy), maximum during one hour.
  Time to laryngeal vestibule opening (LVO, time between tongue tip elevation and pharyngeal phases of swallowing)
Swallowing function- Time to laryngeal vestibule closure (LVC, time between tongue tip elevation and maximal laryngeal closure) | During the ingestion (videofluoroscopy), maximum during one hour.
  Time to laryngeal vestibule closure (LVC, time between tongue tip elevation and maximal laryngeal closure)
Subjective perception of ease of swallowing and oropharyngeal sensation. | Right after ingredient ingestion, maximum during one hour.
  This will be assessed from a questionnaire.

CONTACTS AND LOCATIONS:
Locations (2):
- Grand hopital de Charleroi, Charleroi, Belgium
- Centre Hospitalier Charles Nicolle, Rouen, France

IPD SHARING:
Plan to Share IPD: No